CLINICAL TRIAL: NCT02140307
Title: Study of Potential Health Effects of a Relaxation-response-based Mental Health Promotion Course (RR-MHP) and the Possibilities for Its Applications in the Danish Public Health Sector
Brief Title: Relaxation-Response-based Mental Health Promotion - Open and Calm 2013
Acronym: RR-MHP OC13
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Steen G Hasselbalch (Other)
Collaborators: Nordea-Fonden, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Steen G Hasselbalch, Professor, dr. med., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RR-MHP-OC13
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Stress Psychological; Stress Physiological; Quality of Life
Keywords: Health Promotion; Prevention; Relaxation Response; Meditation; Cortisol
MeSH Terms: conditions — Stress, Psychological | interventions — Calmodulin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Meditation training, group format (Experimental): The course Relaxation Response-based Mental Health Promotion (publicly referred to as "Open and Calm") is given in group format.
  The intervention entails 9 courses (1 per week of 2.5 hrs), a course book (120 pages), audio support (6 guided meditative practices), access to a webpage with additional information, and the possibility of two personal sessions with the intervention instructor (a certified psychologist).
  Interventions: Behavioral: Relaxation Response-based Mental Health Promotion (RR-MHP)
- Meditation training, individual format (Active Comparator): The course Relaxation Response-based Mental Health Promotion ("Open and Calm") is given by the same instructor as for group formats using precisely the same material and methods, but in about 6-9 (as to each persons' individual needs and preferences) face-to-face meetings.
  Interventions: Behavioral: Relaxation Response-based Mental Health Promotion (RR-MHP)
- Wait-list control (No Intervention): This arm is an inactive wait-list control.

INTERVENTIONS:
Behavioral: Relaxation Response-based Mental Health Promotion (RR-MHP) — The Open and Calm intervention is based on a standardized 9-week program. Week 1 uses a simple mantra-based meditation. Week 2 and 5 uses focus on the body. Week 3 and 6 uses focus on thoughts and emotions. Week 4 and 7 uses focus on social relationships. Weeks 8 and 9 were entitled "The focus you feel like", where participants chose their own focus (e.g. two weeks of bodily focus if that was most relevant for a person, while another might chose 1 week focusing on emotions and another focusing on a social relationship).
  Other Names: Open and Calm; Open & Calm; RR-MHP; Relaxation Response Resiliency Program; 3RP
  Arms: Meditation training, group format; Meditation training, individual format

SUMMARY:
The purpose of the study is to investigate health-promoting and stress-reducing psychological, physiological and hormonal effects of a 9-week meditation-based course in personal health and to examine potential baseline factors for any such effects. Thus, the investigators will investigate the course format (individual course or group-based course) as a potential factor the course outcome, and also individual background factors such as demographics and genetic variations.

ELIGIBILITY:
Inclusion Criteria

* Experience of stress, defined as a Cohen's perceived stress scale score > 12.
* Speaks and reads Danish fluently.
* Ability to use the internet to complete questionnaires.
* Participation in face-to-face study information meeting.
* Signed agreement to the study conditions and informed consent form

Exclusion Criteria

* Other current treatment (psychological, medical or other) for stress, depression, anxiety, phobias, traumas or other psychological problems.
* Other current treatment for bodily illnesses, such as pain, migraine, cancer.
* More than one diagnose with psychiatric disease (e.g. anxiety, depression) within the past 3 years.
* Body-Mass Index > 30.
* Major Depression Inventory score > 25 at inclusion interview.
* Physical handicaps affecting life stress or quality of life chronically.
* Drug use (> 50 times hash during the past two years; max 20 times harder drugs, max 2 times per month since the 18th birthday on average; no periods > 3 years where the use of drugs exceeded two times per month).
* Alcohol use > 21 drinks/week for men, and > 14 drinks/week for women and AUDIT-scores (a scale of alcohol-related problems) >20.
* Serious head trauma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Change in scores on Perceived Stress on Cohen's Perceived Stress Scale | From baseline to post-treatment (9 weeks later) and to 3-month follow-up
  The investigators expect a decrease in perceived stress of significantly larger magnitude in interventional groups than in waitlist controls across the three time points
Cortisol secretion as measured by the cortisol awakening response | From baseline to post-treatment (after 9 weeks)
  The investigators expect a significant reduction of cortisol secretion in intervention groups and larger than in wait-list controls. Specifically, the investigators analyze the Area Under Curve with respect to Ground (total cortisol output) after awakening. Cortisol was only collected for 2/3 data waves (N = 48) due to logistics.
  COMMENT: The investigators have two primary outcomes, but both are measures of stress levels. The investigators expect to see both hormonal and perceived stress improvements.

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | From baseline to post-treatment (9 weeks later) and to 3-month follow-up
  The investigators expect a larger improvement of sleep quality in the intervention groups than in the wait-list controls over the course of the three time points
Change in Quality of Life on the WHO-5 scale | From baseline to post-treatment (9 weeks later) and to 3-month follow-up
  The investigators expect a larger improvement in perceived quality of life in intervention groups compared to wait-list controls over the course of the three time points
Change in Short-Form Health Survey-36 | From baseline to post-treatment (9 weeks later) and to 3-month follow-up
  The investigators expect a significantly larger improvement in quality of life (SF-36-Mental Component Summary Score and SF-36 Physical Component Summary Score) in intervention groups compared to wait-list controls over the course of the three time points.
Change in Major Depression Inventory | From baseline to post-treatment (9 weeks later) and to 3-month follow-up
  The investigators expect a significantly larger decrease in depressive symptoms in intervention groups than in wait-list controls over the course of the three time points.

OTHER OUTCOMES:
Changes in physiological stress levels as measured by blood pressure, skin conductance, heart rate variability measures and respiratory measures during resting state (15 minutes). | Baseline to post-treatment (9 weeks)
  The investigators expect larger improvements in intervention groups than in wait-list controls. Due to logistics, only N = 48 were tested physiologically.
Basic processes in visual attention | Baseline to post-treatment (9 weeks)
  The investigators expect larger improvements in intervention groups than wait-list controls for the speed of visual processing (threshold of conscious perception measured in ms) on the Theory of Visual Attention (TVA) task developed at the Center for Visual Cognition, Copenhagen University. The investigators expect a lowered threshold for conscious, visual perception (the TVA-t0 parameter) since they have demonstrated this effect after meditation-based training in a previous study (Jensen et al., 2012, J. Exp. Psych. Gen., MBSR affects Attention)

CONTACTS AND LOCATIONS:
Overall Officials: Christian G Jensen, MSc., Principal Investigator — Neurobiology Research Unit, Copenhagen University Hospital (Rigshospitalet); Steen G Hasselbalch, Professor, Study Director — Memory Clinic, Copenhagen University Hospital (Rigshospitalet); Gitte M Knudsen, Professor, Study Chair — Neurobiology Research Unit, Copenhagen University Hospital (Rigshospitalet)
Locations (1):
- Neurobiology Research Unit, dep. 9201, Copenhagen University Hospital (Rigshospitalet), Copenhagen OE, Denmark

REFERENCES:
- [Derived] Jensen CG, Lansner J, Petersen A, Vangkilde SA, Ringkobing SP, Frokjaer VG, Adamsen D, Knudsen GM, Denninger JW, Hasselbalch SG. Open and Calm--a randomized controlled trial evaluating a public stress reduction program in Denmark. BMC Public Health. 2015 Dec 16;15:1245. doi: 10.1186/s12889-015-2588-2. PMID 26673225
- See also: Homepage of the central investigating research unit — http://www.nru.dk